CLINICAL TRIAL: NCT05660915
Title: A Prospective Clinical Study of the Safety and Efficacy of Robot-assisted Pancreaticoduodenectomy Using an Artery-first Intermediate Approach
Brief Title: A Prospective Clinical Study Using an Artery-first Intermediate Approach in Robot-assisted Pancreaticoduodenectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of University of South China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USC-4310-2
Record Dates: First submitted 2022-11-29; First posted 2022-12-21 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Pancreatic Cancer; Common Bile Duct Diseases; Periampullary Carcinoma
Keywords: Robot-assisted pancreaticoduodenectomy; Superior mesenteric artery first approach; Intermediate approach; Safety and Efficacy; randomized controlled trial
MeSH Terms: conditions — Pancreatic Neoplasms; Common Bile Duct Diseases

STUDY DESIGN:
Intervention Model Description: The key point of surgery in the standard approach group was to first reveal portal vein-superior mesenteric vein and gradually complete the resection of the uncinate process of pancreas based on the reference of portal vein-superior mesenteric vein.In the intermediate approach group, the area between superior mesenteric artery and superior mesenteric vein was defined as the intermediate area and dissection was performed in this area to achieve the removal of the uncinate process of pancreas. Subsequently, data related to intraoperative conditions (such as operation time, amount of blood loss, etc.) and postoperative complications were collected and statistically analyzed to verify the safety of the intermediate approach, and short-term prognostic data was collected to verify its effectiveness.
Who Masked: Outcomes Assessor
Masking Description: The way of surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intermediate approach (Experimental): The key point of surgery in the standard approach group was to first reveal portal vein-superior mesenteric vein and gradually complete the resection of the uncinate process of pancreas based on the reference of portal vein-superior mesenteric vein.
  Interventions: Procedure: Intermediate approach
- The standard approach (Other): The area between superior mesenteric artery and superior mesenteric vein was defined as the intermediate area and dissection was performed in this area to achieve the removal of the uncinate process of pancreas.
  Interventions: Procedure: Standard approach

INTERVENTIONS:
Procedure: Intermediate approach — The area between superior mesenteric vein and superior mesenteric artery was defined as the intermediate area and dissection was performed in this area to achieve the removal of the uncinate process of pancreas.
  Arms: The intermediate approach
Procedure: Standard approach — The key point of surgery in the standard approach group was to first reveal portal vein-superior mesenteric vein and gradually complete the the resection of the uncinate process of pancreas based on the reference of portal vein-superior mesenteric vein.
  Arms: The standard approach

SUMMARY:
Pancreaticoduodenectomy, as a standard surgical procedure for malignant tumors of the head of the pancreas, ampulla and distal common bile duct, has brought the hope of clinical cure for these diseases.In the whole surgical process, the resection of the uncinate process of the pancreas is considered to be a major difficulty in the whole operation, which can affect the rehabilitation process and long-term prognosis. Two main methods have been developed around the dissection of the uncinate process of the pancreas. One is the Venous-first approach based on the portal vein-superior mesenteric vein axis. The other is the Artery-first approach that first explores whether the superior mesenteric artery is invaded by the tumor to judge resectable. The latter is gradually promoted in clinical practice because it can reduce intraoperative bleeding, reduce postoperative complications, and improve long-term prognosis. The intermediate approach is a surgical approach based on the Artery-first approach and adapted to the layout of the robot arm. The area between superior mesenteric artery and superior mesenteric vein was used as an intermediate area to treat the uncinate process of the pancreas in order to reduce perioperative complications and achieve better surgical results. However, the safety and effectiveness of intermediate approach have not been verified,in this prospective clinical study, the investigators will use a robotic surgical platform to perform robot-assisted pancreaticoduodenectomy surgery through the intermediate approach to verify its safety and efficacy.

DETAILED DESCRIPTION:
Firstly, according to the inclusion and exclusion criteria, all patients from the First Affiliated Hospital of the University of South China who were to undergo robot-assisted pancreaticoduodenectomy were randomized into two groups, namely the standard approach group and the intermediate approach group. The two groups were under the management of the same surgical team throughout the perioperative period, and were managed according to standardized Enhanced recovery after surgery approach. The brief procedure includes: (1) Placement of the trocar in appropriate place; (2) An ultrasonic knife was used to cut the appetizing colonic ligament and expose the pancreas. The superior mesenteric vein, common hepatic artery, proper hepatic artery and gastroduodenal artery were exposed, and the adjacent lymph nodes were dissected. The right gastric artery and gastroduodenal artery were resected to expose the portal vein. Dissect the common bile duct and peel the gallbladder from the bile fossa; The free common bile duct was dissected and suspended with a vascular sling. (3) Resection of distal stomach and jejunum. The pancreas was cut off with ultrasonic knife. (4) Child reconstruction - pancreaticojejunostomy (pancreatic duct to jejunal mucosa anastomosis) , cholangiojejunostomy and gastrojejunostomy were adopted. (5) Thoroughly rinse the abdominal cavity and place the abdominal drainage tube properly after checking for no active bleeding.The key point of surgery in the standard approach group was to first reveal portal vein-superior mesenteric vein and gradually complete the resection of the uncinate process of pancreas based on the reference of portal vein-superior mesenteric vein. In the intermediate approach group, the area between superior mesenteric vein and superior mesenteric artery was defined as the intermediate area and dissection was performed in this area to achieve the removal of the uncinate process of pancreas. Subsequently, data related to intraoperative conditions (such as operation time, amount of blood loss, etc.) and postoperative complications were collected and statistically analyzed to verify the safety of the intermediate approach, and short-term prognostic data was collected to verify its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Preoperative imaging suggested the presence of space occupying in the head of the pancreas, ampullary abdomen, and distal common bile duct tumor lesions to be treated with Pancreaticoduodenectomy
* No obvious arterial invasion, no obvious venous invasion or vein invasion but can be replaced
* No distant transfer
* Complete clinical data

Exclusion Criteria:

* With tumors of other organs
* Patients unable to tolerate anesthesia and operation due to serious abnormalities in functions of heart, lung and other important organs
* Patients found intraoperative peripheral organ metastasis combined with excision of other organs or found intraoperative radical excision could not be performed and underwent palliative drainage surgery or end the surgery
* Preoperative adjuvant therapy was given
* Clinical data are seriously missing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Rate of mortality after surgery | 5 months
  The short-term prognosis of this procedure will be evaluated by recording patient mortality during hospitalization, 30 days and 90 days after surgery.

SECONDARY OUTCOMES:
Unplanned re-admission rate after discharge within 30 days | 3 months
  Serious discomfort requiring re-admission within 30 days after discharge will be recorded, and the safety of the surgical method will be evaluated by this indicator.
Incidence of postoperative complications | 2 months
  During hospitalization, common complications of pancreaticoduodenectomy, such as postoperative pancreatic fistula, bile leak, gastrojejunostomy leak, and delayed gastric emptying, will be recorded according to the international diagnostic criteria to evaluate the short-term safety of this surgical approach.

CONTACTS AND LOCATIONS:
Overall Officials: Guodong Chen, PhD, Study Chair — The First Affiliated Hospital of University of South China
Locations (1):
- The First Affiliated Hospital of University of South China, Hengyang, Hunan, China

IPD SHARING:
Plan to Share IPD: No